CLINICAL TRIAL: NCT03593304
Title: Randomized, Double-blind, Placebo Controlled, Multicenter Trial to Evaluate the Neuroprotective Effect of Vitamin B6 and Vitamin B12 Against Vincristine Induced Neurotoxicity in Acute Lymphoblastic Leukaemia Patients
Brief Title: Evaluate the Neuroprotective Effect of Vitamin B6 and Vitamin B12 Against Vincristine Induced Neurotoxicity in Acute Lymphoblastic Leukaemia Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Ferdaush Ahmed Sojib, Resident, Department of Pharmacology, BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: No. BSMMU/2018/2105
Record Dates: First submitted 2018-03-10; First posted 2018-07-20 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Vincristine Induced Neurotoxicity; Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vitamin B 12; Vitamin B 6; Saline Solution; Pyridoxine

STUDY DESIGN:
Intervention Model Description: Experimental group: Medicine- Injection Mecobalamin (500mcg), Tablet Pyridoxine hydrochloride (25 mg) Placebo group: Injection normal saline (1ml), oral placebo pill
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Mecobalamin and Pyridoxine hydrochloride (Active Comparator): Injection Mecobalamin (500mcg) three times a week (on day 1,3,5 of vincristine chemotherapy) for 5 weeks.Tablet Pyridoxine hydrochloride (25 mg) 2 tablets thrice daily for 5 weeks.
  Interventions: Drug: Injection Mecobalamin; Drug: Tablet Pyridoxine hydrochlorid
- Placebo: normal saline and Oral placebo (Placebo Comparator): Injection normal saline (1ml) three times a week (on day 1,3,5 of vincristine chemotherapy) for 5 weeks.Oral placebo pill 2 tablets thrice daily for 5 weeks.
  Interventions: Drug: Normal saline; Drug: Oral Placebo

INTERVENTIONS:
Drug: Injection Mecobalamin — Injection Mecobalamin (500mcg) three times a week (on day 1,3,5 of vincristine chemotherapy) for 5 weeks.
  Other Names: Vitamin B12
  Arms: Experimental:Mecobalamin and Pyridoxine hydrochloride
Drug: Tablet Pyridoxine hydrochlorid — Tablet Pyridoxine hydrochloride (25 mg) 2 tablets thrice daily for 5 weeks.
  Other Names: Vitamin B6
  Arms: Experimental:Mecobalamin and Pyridoxine hydrochloride
Drug: Normal saline — Injection Normal saline(1ml) three times a week (on day 1,3,5 of vincristine chemotherapy) for 5 weeks.
  Other Names: Placebo for mcobalamin
  Arms: Placebo: normal saline and Oral placebo
Drug: Oral Placebo — Placebo Oral Tablet (25 mg) 2 tablets thrice daily for 5 weeks.
  Other Names: Placebo for pyridoxine hydrochloride
  Arms: Placebo: normal saline and Oral placebo

SUMMARY:
This study will be conducted to evaluate the effect of vitamin B6 and vitamin B12 in reducing the incidence and severity and delaying the onset of Vincristine Induced neurotoxicity in Acute Lymphobalstic Leukemia (ALL) patient.

DETAILED DESCRIPTION:
Acute lymphoblastic leukaemia (ALL) is increasing day by day in less developed countries like Bangladesh. Vincristine is one of the important chemotherapeutic agents used in combination with other medicines to treat Acute Lymphoblastic Leukemia (ALL). Good prognostic outcome of ALL depends on uninterrupted and complete course of chemotherapy. With full course of treatment about 85% of adult patients and 98% of children attain complete recovery. Development of some deleterious adverse effects especially neurotoxicity results in dose reduction, protocol deviation and even abandonment of treatment. About 45% patients develop peripheral neuropathy and more than 33% patients develop autonomic neuropathy who needs dose reduction or treatment protocol deviation. Many studies have been conducted to explore the potential of medicine to prevent or treat neuropathy but still there is no success. This proposed study will be an effort to identify the potential of vitamin B6 (Pyridoxine hydrochloride) and vitamin B12 (Mecobalamin) as preventive measure in reducing the incidence, risk, severity and time of onset of vincristine induced neurotoxicity. This study will be a multicenter, double blind, randomized controlled trial. In this study newly diagnosed ALL patients will be enrolled in induction phase and patients will be randomly allocated into two arms by using online graph pad software. After assessing the baseline characteristics by Eastern Cooperative Oncology Group (ECOG) performance status and Composite Autonomic Symptom Score (COMPASS 31), patient will be provided medicine or placebo. From the day of starting chemotherapy, patients on intervention arm will be administered vitamin B6 and vitamin B12. Vitamin B6 will be given 50 mg thrice daily orally for 5 weeks and Vitamin B12 will be given 500 μg three times weekly intravenously on day 1, 3 and 5 of every week for 5 weeks. On the other hand, patients on placebo arm will be given placebo pill and injection at same interval. Each patient will be evaluated for neurotoxicity on the outset of every 2nd, 3rd, 4th and 5th week by using COMPASS 31 for autonomic neuropathy. Incidence, severity and onset will be compared on both arms. After approval from institutional review board (IRB) every eligible patient will be informed about the intervention and the study. Informed written consent will be taken of the patients who will take part in the study willingly. Patient's anonymity will be maintained and will be used for research purpose only.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older with newly diagnosed ALL going to start induction chemotherapy with Vincristine
* Patients ECOG Performance Status 0 to 3
* Patients with no preexisting autonomic neuropathy
* Patients with normal renal function (Serum creatinine <1.5 mg/dl)
* No history of diabetes mellitus
* Patients agree to participate in the study signing an informed written consent

Exclusion Criteria:

* Pregnant women and nursing mothers
* Patients with clinical neuropathy due to diabetes mellitus and other causes like multiple sclerosis, spinal cord injury, post stroke
* Patients with head neck tumors
* Patients taking anticonvulsants, antidepressants, opioids, vitamin E and other neuropathic pain medication agents like topical anesthetic agents, non steroidal anti-inflammatory drugs (NSAIDs)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Vincristine Induced neurotoxicity | Cumulative incidence at 5th week of vincristine chemotherapy
Severity of Vincristine Induced neurotoxicity | On the outset of 1st week change in the severity of neurotoxicity on the outset of 2nd week, 3rd week, 4th week, 5th week of vincristine chemotherapy
  Changes of severity will be assessed by COMPASS 31 on the outset of 2nd week, 3rd week, 4th week, 5th week of vincristine chemotherapy
Time of onset of Vincristine Induced Neurotoxicity | 1st week (baseline), change in neurotoxicity status on the outset 2nd week, 3rd week, 4th week and 5th week of vincristine chemotherapy
  change in neurotoxicity status on the outset of 2nd week, 3rd week, 4th week, 5th week of vincristine chemotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Bangabandhu Sheikh Mujib Medical University, Dhaka, Shahbag
  - Dhaka Medical College Hospital, Dhaka